CLINICAL TRIAL: NCT05918237
Title: Pilot Study to Test the Effects of Arctiva on Mild to Moderate Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ClinOhio Research Services, LLC (Industry)
Collaborators: Arctiva Wellness LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECZPROTOCOLOHIO115
Record Dates: First submitted 2023-06-14; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Atopic Dermatitis Eczema

STUDY DESIGN:
Intervention Model Description: Open label, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Arctiva — A colloidal oatmeal cream designed to stimulate healing and repair of damaged tissue naturally, working with the body instead of against it.

SUMMARY:
Up to 30 participants with mild to moderate atopic dermatitis/eczema will be enrolled to apply study Investigational Product for 4 weeks.

DETAILED DESCRIPTION:
This will be a 4-week single arm study. This study will be executed by one clinical research company in one research center accruing 30 subjects with mild to moderate Eczema/atopic dermatitis. Patients ages 18-75, will be enrolled. Subjects that are enrolled will be placed on Locus's Over The Counter cream "Arctiva" twice per day for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female;18-75 years of age
* Have a clinical diagnosis of Mild to Moderate Eczema or Atopic Dermatitis
* Signed and dated written informed consent in accordance with Good Clinical Practice (GCP) and local legislation prior to the start of any screening procedure

Exclusion Criteria:

* Patients using topical corticosteroids steroidal creams and other agents within 7 days prior to first dose of trial Eczema treatment.
* Use of systemic corticosteroids or other agents for atopic dermatitis within 4 weeks prior to first dose of trial treatment.
* Active bacterial, viral, or fungal skin infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Severity Scoring of Atopic Dermatitis Index (SCORAD) improvement [Timeframe : Baseline to Day 28] | 28 Days
  Change from Baseline to Day 28 in overall Severity Scoring of Atopic Dermatitis Index (SCORAD)

SECONDARY OUTCOMES:
Change from Baseline in Dermatology Life Quality Index (DLQI) [Timeframe: Baseline to Day 28] | 28 Days
  Change from baseline to Day 28 in Dermatology Life Quality Index (DLQI) evaluating the impact on Quality of life scale: Very much ; A lot; a little or Not at all.
Change from baseline in Patient-Oriented Eczema Measure (POEM). [ Time Frame: Baseline and 28 Days] | 28 Days
  Change from baseline to Day 28 in Patient-Oriented Eczema Measure (POEM) investigating the number of days patients have been subjected, due to eczema, to itchy skin, sleep disturbance; skin bleeding; skin weeping; skin cracked; skin flaking and skin dryness. Scale defined as : 0 = no days; 1= 1-2 days; 2= 3-4 days; 3= 5-6 days; 4 = everyday

CONTACTS AND LOCATIONS:
Locations (1):
- ClinOhio Research Services, LLC, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No